CLINICAL TRIAL: NCT00316316
Title: Cognitive Behavioral Therapy Plus Motivational Interviewing for Obsessive Compulsive Disorder
Brief Title: Cognitive Behavioral Therapy Plus Motivational Interviewing for Treatment of Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #5124; R34MH071570 (NIH); DAHBR 96-BHA
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Participants will receive motivational interviewing plus exposure and response prevention
  Interventions: Behavioral: Motivational interviewing plus exposure and response prevention (MI plus EX/RP)
- 2 (Active Comparator): Participants will receive exposure and response prevention only
  Interventions: Behavioral: Exposure and response prevention (EX/RP)

INTERVENTIONS:
Behavioral: Motivational interviewing plus exposure and response prevention (MI plus EX/RP) — Participants will receive 18 sessions of MI plus EX/RP.
  Other Names: MI plus EX/RP
  Arms: 1
Behavioral: Exposure and response prevention (EX/RP) — Participants will receive 18 sessions of EX/RP.
  Other Names: EX/RP
  Arms: 2

SUMMARY:
This study will determine the effectiveness of adding motivational interviewing to cognitive behavioral therapy, consisting of exposure and ritual prevention, in improving treatment outcomes in people with obsessive-compulsive disorder.

DETAILED DESCRIPTION:
Obsessive Compulsive Disorder (OCD) is a chronic and debilitating anxiety disorder. People with OCD often experience recurrent unwanted thoughts, or obsessions. Some examples of obsessions include the following: repetitive fears of causing harm or being harmed; fears of contamination and illness; fears of making mistakes; intrusive distressing sexual or religious imagery; and fears of losing things. In an effort to relieve anxiety about these obsessions, people with OCD develop repetitive behaviors called compulsions. Some examples of compulsions include the following: repetitive washing and cleaning; excessive checking; excessive ordering and arranging; and extreme hoarding and saving. These thoughts and behaviors interfere with everyday life to a great extent. Cognitive behavior therapy (CBT) with exposure and ritual prevention (EX/RP) is a standard treatment for OCD. EX/RP involves both imaginary and real exposure to situations or settings that may stimulate OCD behavior, and it requires that patients refrain from ritualizing. Motivational interviewing (MI) may help to enhance an individual's motivation to change by exploring and resolving ambivalence. This study will determine the effectiveness of adding MI to CBT that consists of EX/RP in improving treatment outcome in people with OCD.

Participants in this single-blind study will be randomly assigned to receive either standard CBT with EX/RP or CBT with EX/RP plus MI. All participants will report to the study site twice weekly for both therapy and assessments for a total of 2 months. Assessments will include interviews and self-rating forms. No medication will be administered during this study. However, participants will continue on any medication that they are taking at the time of study entry. All participants will be assessed for outcomes upon study completion. Participants who respond to therapy will be assessed again 6 months following study completion.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of OCD as defined by DSM-IV
* Obsessions and/or compulsions must have been present for at least one year
* At pre-treatment, a minimum on Y-BOCS on items 1-10 of 16
* If on psychiatric medication, patient has been on stable SRI dose for a minimum of 12 weeks (and four weeks for concomitant OCD meds,e.g., benzos and antipsychotics) and plans to remain on a stable dose for the duration of the EX/RP+MI treatment.
* Able to provide informed consent
* No prior adequate EX/RP treatment (defined as at least 8 exposure sessions that include response prevention instructions and between sessions assignments in a 2 month period)
* Based on hx, subject is unlikely to require a change in med during the course of EX/RP/EX/RP+MI treatment

Exclusion Criteria:

* Any additional medical or psychiatric conditions that could make participation in the study medically inadvisable
* Currently receiving psychotherapy at another clinic

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Obsessive-compulsive symptoms | Measured at Months 2 and 8

SECONDARY OUTCOMES:
Adherence, depression, insight, and quality of life | Measured at Months 2 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Helen Blair Simpson, MD, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Farris SG, McLean CP, Van Meter PE, Simpson HB, Foa EB. Treatment response, symptom remission, and wellness in obsessive-compulsive disorder. J Clin Psychiatry. 2013 Jul;74(7):685-90. doi: 10.4088/JCP.12m07789. PMID 23945445
- See also: Click here for the Obsessive-Compulsive Disorder Research Clinic website. — http://www.Columbia-OCD.org